CLINICAL TRIAL: NCT02089958
Title: Standardization of Laparoscopic Intraperitoneal Onlay Mesh Augmentation for Incisional Hernia Repair: Impact on Clinical Outcomes and Quality-of-Life - Open Prospective Observational Multicentre Cohort Study
Brief Title: Standardization of Laparoscopic Hernia Repair
Acronym: LIPOM
Status: Completed | Type: Observational
Sponsor: Klinikum Fulda (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Achim Hellinger, Priv. Doz. Dr. med., Klinikum Fulda
Other Study IDs: AE 003
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Incisional Hernia
Keywords: Lapraoscopy, incisional hernia repair, mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laparoscopic incisional hernia repair: Incisional hernia, LIPOM
  Interventions: Procedure: Laparoscopic incisional hernia repair

INTERVENTIONS:
Procedure: Laparoscopic incisional hernia repair — Standardized laparoscopic incisional hernia repair with mesh
  Other Names: LIPOM

SUMMARY:
Incisional hernias are one of the most frequent complications in abdominal surgery. Laparoscopic repair is widely used but even not standardized. Existing data from different study designs show no representative data resulting in a lack of comparability and evidence. Therefore the standardization of operative techique has been proposed by the LIPOM-study group and will be assessed in a prospective manner.

DETAILED DESCRIPTION:
Data are scheduled for publication.

ELIGIBILITY:
Inclusion Criteria:

* Primary incisional hernia
* Hernia size EHS W 1-2
* Hernia location EHS M 1-5, L 1-3
* Clinical symptoms or progressive growth of hernia

Exclusion Criteria:

* Recurrent incisional hernia
* Ventral hernie
* Hernia size > EHS W 2
* Hernia location EHS L 4, ASA >3
* Prospective mesh overlap < 5 cm
* Malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pts. with incisional hernia following prior abdominal surgery
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | until 12 mths postoperatively

SECONDARY OUTCOMES:
Pain, Quality of Life | until 12 mths postoperatively
  Pain measured by numeric rating scale. QoL measured by Carolina Comfort Scale.

OTHER OUTCOMES:
Wound infection | 12 mts postoperatively
  Measured along SSI-classification

CONTACTS AND LOCATIONS:
Overall Officials: Achim Hellinger, MD, PhD, Study Chair — Klinikum Fulda
Locations (1):
- Klinikum Fulda, Fulda, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Derived] Hellinger A, Wotzlaw F, Fackeldey V, Pistorius G, Zdichavsky M, Junemann R, Buia A. Development of an open prospective observational multicentre cohort study to determine the impact of standardization of laparoscopic intraperitoneal onlay mesh repair (IPOM) for incisional hernia on clinical outcome and quality of life (LIPOM-Trial). Contemp Clin Trials Commun. 2016 Aug 11;4:118-123. doi: 10.1016/j.conctc.2016.08.001. eCollection 2016 Dec 15. PMID 29736474